CLINICAL TRIAL: NCT04606147
Title: Comparison of Effectiveness of Ultrasound Guided Erector Spinae Plane Block With Ultrasound Guided Serratus Anterior Block in Modified Radical Mastectomy, Randomized Single Blinded Comparative Study.
Brief Title: Effectiveness of Ultrasound Guided Erector Spinae Plane Block Against Ultrasound Guided Serratus Anterior Block in Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mohammed Magdy Abdelrahman Elsayed, Resident of Anaesthesiology, ICU and Pain Management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MS-268-2019
Record Dates: First submitted 2020-10-21; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer; Postoperative Pain
Keywords: Modified Radical Mastectomy MRM, ESPB ,SAPB , Regional anesthesia and postoperative analgesia.
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Performer of nerve blocks will know type of block but investigator for postoperative pain will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 ((Serratus Anterior Plane Block SAPB)) N=3o (Experimental): Patients received Ultrasound guided Serratus Anterior Plane Block preoperative with injection of 30 ml levobupivacaine 0.25%. Then patients were transferred to the operating room.
  Interventions: Procedure: Serratus Anterior Plane Block
- Group 2 ((Erector Spinae Plane Block ESPB)) N=3o (Experimental): Patients received Ultrasound guided erector spinae plane block with injection of 30 ml levobupivacaine 0.25%. Then patients were transferred to the operating room.
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Serratus Anterior Plane Block — The block is performed with full aseptic precautions.in lateral position &arm abduction. US probe placed on the patient's midaxillary line in the transverse plane, at the level of the fifth rib.With the rib, pleural line, and overlying serratus anterior and latissimus dorsi muscles visualized, the skin and subcutaneous tissue can be topicalized. Then, using ultrasound guidance, A regional block needle is advanced in-plane at an angle of approximately 45 degrees towards the fifth rib.Correct location of the needle tip in the fascial plane deep to serratus anterior muscle will be confirmed by injecting 0.5-1 ml normal saline and seeing hydrodissection of fascial plane between SAM and 5th rib. After aspiration to avoid intravascular injection 30 ml of levobupivacaine 0.25% is injected anteriorly to the rib and deep to the serratus anterior muscle. The entirety of the needle should be visualized at all times throughout the procedure.
  Arms: Group 1 ((Serratus Anterior Plane Block SAPB)) N=3o
Procedure: Erector spinae plane block — The block is performed with full aseptic precautions at T5 level. T5 transverse process is identified by us as flat, squared-off acoustic shadows with only a very faint image of the pleura.In longitudinal us view following layers will be visible superficial to transverse processes: skin and subcutaneous tissue, trapezius, erector spinae muscle.Skin is topicalised , then echogenic block needle inserted in- plane to the ultrasound beam in a cranial-to-caudal direction until contact is made with the T5 transverse process. After aspiration to avoid intravascular injection 30 ml levobupivacaine 0.25% was injected and separation was seen. 6-13-MHz, linear transducer set for small parts and a depth of 4-6 cm was used
  Arms: Group 2 ((Erector Spinae Plane Block ESPB)) N=3o

SUMMARY:
The aim of this study is to compare and evaluate the safety and analgesic efficacy of ultrasound guided ESP block and ultrasound guided serratus anterior plane block in patients undergoing modified radical mastectomy.

DETAILED DESCRIPTION:
Methodology:

This Randomised Comparative Single Blinded Study was conducted at National Cancer Institute Cairo University after approval by the institutional review board, scientific committee of Anesthesia department Kasr Alainy Cairo University (02/10/2019 Code: N - 65\2019 ms) and Ethical committee at Kasr Alainy Cairo University (1\ 12 \2019 code: MS-268-2019)

Type of consent of study participants: Written and verbal

Study Methods:

Population of study: 60 Female patients ASA II, III scheduled for modified radical mastectomy under general anaesthesia.

Methodology in details:

Randomization:

The patients were randomly assigned into two equal comparable groups using computer- generated random numbers in opaque closed envelopes, each of which included 30 patients.

Randomization was done by a statistician and group of the patient was revealed only when the included patient is transferred to the preanesthetic room.

Study Protocol:

Patient assessment; History, physical exam, laboratory and radiological investigations at preoperative assessment clinic National Cancer Institute Cairo University.

Preoperative assessment at night of surgery. The patients were instructed how to report pain by means of Numeric Pain Rating Scale, in which 0 = no pain and 10 =worst possible pain. Informed consent was obtained.

Preoperative fasting; minimum of 6 hours for food and minimum of 2 hours for water and clear fluids. 20G IV cannula was inserted. All patients premedicated with IV midazolam 0.01-0.02mg\kg 30 minutes preoperatively. Both blocks were done preoperative with the patients at lateral position.

After allocation of the patient to a study group patients of group 1 received serratus anterior plane block and patients of group 2 received erector spinae plane block.

Serratus Anterior Plane Block Technique;

The block is performed with full aseptic precautions. Lateral Decubitus with arm abduction is preferred. Ultrasound probe should be placed on the patient's midaxillary line in the transverse plane, at the level of the fifth rib, with the indicator oriented toward the operator's left. With the rib, pleural line, and overlying serratus anterior and latissimus dorsi muscles visualized, the skin and subcutaneous tissue can be topicalized with 3 ml of lidocaine 1%. Then, using ultrasound guidance, A 38-mm 22-gauge regional block needle is advanced in-plane at an angle of approximately 45 degrees towards the fifth rib.

Correct location of the needle tip in the fascial plane deep to serratus anterior muscle will be confirmed by injecting 0.5-1 ml normal saline and seeing hydrodissection of fascial plane between SAM and 5th rib. After aspiration to avoid intravascular injection 30 ml of levobupivacaine 0.25% is injected anteriorly to the rib and deep to the serratus anterior muscle. The entirety of the needle should be visualized at all times throughout the procedure, and care should be taken to avoid any vessels while traversing the soft tissue.6-13-MHz, linear transducer set for small parts and a depth of 1-4 cm was used for this block.

Erector spinae plane block Technique; The block is performed with full aseptic precautions. Block level at T5. Ultrasound probe placed on the back in a transverse orientation to identify the tip of the T5 transverse process; these are recognizable as flat, squared-off acoustic shadows with only a very faint image of the pleura visible. If the transducer is too lateral, the ribs will be visualized instead; these are recognizable as rounded acoustic shadows with an intervening hyperechoic pleural line. The tip of the transverse process centered on the ultrasound screen and the probe will then be rotated into a longitudinal orientation to produce a parasagittal view, in which the following layers will be visible superficial to the acoustic shadows of the transverse processes: skin and subcutaneous tissue, trapezius, erector spinae muscle and T5 transverse process. A skin wheal using 3ml of 1% lidocaine is made , then echogenic block needle will be inserted in- plane to the ultrasound beam in a cranial-to-caudal direction until contact is made with the T5 transverse process. Correct location of the needle tip in the fascial plane deep to erector spinae muscle will be confirmed by injecting 0.5-1 ml normal saline and seeing the fluid lifting the erector spinae muscle off the transverse process without distending the muscle. After aspiration to avoid intravascular injection 30 ml levobupivacaine 0.25% was injected and separation was seen. 6-13-MHz, linear transducer set for small parts and a depth of 4-6 cm was used (59-62).

In both blocks Fujifilm Sonosite M-Turbo Ultrasound system was used.

After performing blocks lung ultrasound was performed to exclude pneumothorax, chest was divided to 6 quadrants with the patient semi sitting:

Anterior upper and lower quadrants Lateral upper and lower quadrants Posterior upper and lower quadrants All quadrants scanned especially upper quadrants was scanned looking for signs of pneumothorax such as absence of lung sliding, presence of B lines, barcode or stratosphere sign and lung-point sign. 6-13-MHz, linear transducer set for small parts and a depth of 4-6 cm was used.

Lung us was done after performing block and post operative at PACU

Patients transferred to the post-anaesthesia care unit (PACU) where the Numeric Pain Rating Scale score, MAP and heart rate were noted immediately on arrival, where they will be observed for 2 hours then discharged to the ward. Lung ultrasound was done once again at PACU looking for signs of pneumothorax. Rescue analgesia was provided in the form of IV morphine 3 mg boluses when the patient indicates Numeric Pain Rating Scale score ≥ 4. The total amount of morphine given in 24 hours was recorded for the two groups. A maximum dose of 0.5 mg/kg/24hours of morphine was allowed.

After that Modified Radical Mastectomy is performed under GA.

After the patients were transferred to their respective ward, Multimodal analgesia was provided as the following:

IV paracetamol 500 mg \6 hours IV ketorolac 30mg\8 hours.

Sample size:

The investigators plan was to study continuous response variable (post operative morphine consumption in the1 st 24 hours) from independent control and experimental with 1 control per 1 experimental subject. The experimental group is Erector spinae plane block (ESPB) versus control group Serratus Anterior Plane Block (SAP). In a previous randomized controlled trial by Gupta et al (2017), comparing Analgesic efficacy of ultrasound-guided paravertebral block with serratus anterior plane block for modified radical mastectomy mean postoperative morphine consumptions in (SAP) group was found to be 9.2 ± 2.1 mg. In another study by Singh et al (2019), which compares analgesic efficacy of Erector spinae plane block (ESPB) with opioid based anaesthesia mean postoperative morphine consumptions in (ESPB) was 1.9 ± 2.01 mg. If the true difference in the control and experimental means is7.8, A sample size of 14 experimental subjects and 14 control subjects was needed to be able to reject the null hypothesis that the experimental and control groups are equal with probability(power) of 0.9. Type 1 error probability associated with this test of this null hypothesis is 0.01. To ensure normal distribution of response variables 30 patients per group were recruited.

Statistical analysis:

SPSS version 23.0 was used in data analysis. Mean and standard deviation described quantitative data with median and range when appropriate. Quantitative variables were tested for normality to select appropriate statistical tests. Comparison of means (or medians) of two independent groups was done using t test (parametric or non- parametric). To show the effect of time on vitals, parametric repeated measures ANOVA (or non-parametric Friedman tests) were used to show changes overtime both intra and post-operative. Post-hoc test were used for pairwise comparisons and were Bonferroni adjusted. Chi-square and Fisher Exact were used for testing proportion independence. P value was always two tailed and set significant at 0.05 level.

Sources of funding: National Cancer Institute Cairo University No conflict of interest.

ELIGIBILITY:
Inclusion criteria:

* Female patients
* Type of surgery; Modified Radical Mastectomy MRM
* Physical status ASA II, III.
* Age ≥ 18 and ≤ 65 Years.
* Body mass index (BMI): ≥ 20 kg/m2 and ≤ 35 kg/m2.

Exclusion criteria:

* Age: ≤18 years or ≥65 years
* BMI: ≤20 kg/m2 or ≥ 35 kg/m2
* Known sensitivity or contraindication to drugs used in the study (local anaesthetics, opioids).
* History of psychological disorders and/or chronic pain syndrome.
* Contraindication to regional anaesthesia e.g. local sepsis, pre-existing peripheral neuropathies and coagulopathy.
* Patient refusal.
* Severe respiratory or cardiac disorders.
* Advanced liver or kidney disease.
* Pregnancy.
* Physical status ASA IV
* Male patients.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Total amount of postoperative morphine consumption in 24 hours. (mg) | 24 hours
  Total amount of postoperative morphine consumption in 24 hours. (mg)

SECONDARY OUTCOMES:
Total amount of intraoperative fentanyl consumption (mcg) | duration of surgery
  Total amount of intraoperative fentanyl consumption (mcg)
Change in heart rate intraoperatively | duration of surgery
  Introperative measurement of HR at 30 minutes interval in comparison to baseline reading.
The degree of postoperative sedation according to Ramsay scores. | 24 hours
  Post operative sedation according to Ramsay scores at 0,2,4,8,12,16,20,24 hours:
  (1 = anxious or restless or both; 2 = cooperative, orientated, and tranquil; 3= responding to commands; 4 = brisk response to stimulus; 5 = sluggish response to stimulus; and 6 = no response to stimulus). A Ramsay score of 5 or 6 considered excessively high sedation levels; a Ramsay score of 2 to 4 considered adequate sedation levels needing observation; a Ramsay score of 1 considered inadequate or insufficient sedation Levels.
Time to first rescue analgesia (hours) | postoperative
  duration of analgesic effect until the time of 1st rescue analgesia
Numeric Pain Rating Scale score, both at rest and during movement | 24 hours
  Numeric Pain Rating Scale score, both at rest and during movement at PACU, and every 4 hours until 24 hours postoperatively.The patients were instructed how to report pain by means of Numeric Pain Rating Scale, in which 0 = no pain and 10 =worst possible pain.
Block related complications | 24 hours
  Complications related to blocks such as local anaesthetic systemic toxicity, pneumothorax and arterial puncture.
Patient satisfaction | 24 hours
  the patients will be classified in this group to: satisfied or not.
Change in mean arterial blood pressure intraoperatively | duration of surgery
  ntroperative measurement of MAP at 30 minutes interval in comparison to baseline reading.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed I Hammimy, Professor, Study Chair — Anaesthesiology Faculty of Medicine - Cairo University; Ahmed F Zaghlol, Assistant Professor, Study Director — Anaesthesiology Faculty of Medicine - Cairo University; Fatima A El Shamy, Lecturer, Study Director — Anaesthesiology National Cancer Institute - Cairo University; Mohhamed M Abdelrahman, M.B. B.CH, Principal Investigator — Anaesthesiology National Cancer Institute - Cairo University
Locations (1):
- National Cancer Institute - Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Garg R, Bhan S, Vig S. Newer regional analgesia interventions (fascial plane blocks) for breast surgeries: Review of literature. Indian J Anaesth. 2018 Apr;62(4):254-262. doi: 10.4103/ija.IJA_46_18. PMID 29720750
- [Background] De Cassai A, Bonvicini D, Correale C, Sandei L, Tulgar S, Tonetti T. Erector spinae plane block: a systematic qualitative review. Minerva Anestesiol. 2019 Mar;85(3):308-319. doi: 10.23736/S0375-9393.18.13341-4. Epub 2019 Jan 4. PMID 30621377
- [Background] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Background] Smith WC, Bourne D, Squair J, Phillips DO, Chambers WA. A retrospective cohort study of post mastectomy pain syndrome. Pain. 1999 Oct;83(1):91-5. doi: 10.1016/s0304-3959(99)00076-7. PMID 10506676
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Gupta K, Srikanth K, Girdhar KK, Chan V. Analgesic efficacy of ultrasound-guided paravertebral block versus serratus plane block for modified radical mastectomy: A randomised, controlled trial. Indian J Anaesth. 2017 May;61(5):381-386. doi: 10.4103/ija.IJA_62_17. PMID 28584346
- [Background] Singh S, Kumar G, Akhileshwar. Ultrasound-guided erector spinae plane block for postoperative analgesia in modified radical mastectomy: A randomised control study. Indian J Anaesth. 2019 Mar;63(3):200-204. doi: 10.4103/ija.IJA_758_18. PMID 30988534